CLINICAL TRIAL: NCT05039684
Title: Inflammatory Biomarkers in Ocular Surface in Patients With Primary Open Angle Glaucoma and Ocular Hypertension Under Topical Prostaglandin Therapy
Brief Title: Inflammatory Biomarkers in Ocular Surface in Primary Open Angle Glaucoma or Ocular Hypertension Under Topical Prostaglandins
Status: Recruiting | Type: Observational
Sponsor: Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other)
Collaborators: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Sponsor
Other Study IDs: IOBA-2021-44
Record Dates: First submitted 2021-08-27; First posted 2021-09-09 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
Keywords: glaucoma; prostaglandin; ocular hypertension; biomarker; inflammation; confocal in-vivo microscopy; cornea; tear film; conjunctiva; impression cytology
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma; Inflammation; Corneal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — A 1-2 microL tear sample. Conjunctival impression cytology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Primary open angle glaucoma / ocular hypertension - Treatment with Xalatan: Patients with primary open angle glaucoma or ocular hypertension treated with Xalatan
- Primary open angle glaucoma / ocular hypertension - Treatment with Monoprost: Patients with primary open angle glaucoma or ocular hypertension treated with Monoprost
- Primary open angle glaucoma / ocular hypertension - Treatment with Saflutan: Patients with primary open angle glaucoma or ocular hypertension treated with Saflutan
- Ocular hypertension - No treatment: Patients ocular hypertension untreated

SUMMARY:
Glaucoma is a chronic optic neuropathy whose main modifiable risk factor is an abnormally elevated intraocular pressure. The aim of glaucoma treatment is to slow the progression of the disease by reducing intraocular pressure.

Prostaglandin derivatives are the most effective topical drugs in reducing intraocular pressure (IOP). Among these, latanoprost was the first agent of this type to be approved for use in patients with glaucoma or ocular hypertension.

These eye drops are available with and without preservatives. There are two commercial brands in our environment, Xalatan®, which contains 0.005% latanoprost and 0.2 mg/ml benzalkonium chloride (BAK) and Monoprost®, which contains the same amount of latanoprost but does not carry a preservative. The prostaglandin analog with a lower concentration of active ingredient available in Spain without preservative is tafluprost 0.0015%, commercially available under the name Saflutan®.

The long-term use of hypotensive eye drops with preservatives generates changes in the ocular surface, such as instability of the tear film, conjunctival inflammation, subconjunctival fibrosis, apoptosis of the conjunctival epithelium and deterioration of the corneal surface, causing symptoms such as stinging, tearing, sensation foreign body, photophobia and blurred vision.

This research will evaluate the changes in the ocular surface and in the expression of inflammatory molecules that occur in the conjunctiva in patients with a diagnosis of glaucoma and ocular hypertension who are under ocular hypotensive treatment with tafluprost, comparing it with the two commercial preparations of latanoprost.

These three groups of patients will have a control group of patients with a diagnosis of ocular hypertension who will not have any topical hypotensive medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary open angle glaucoma or ocular hypertension as defined in Early Manifest Glaucoma Trial
* > 18 years old
* Signed informed consent
* 3 or more months under monotherapy treatment with tafluprost 0.0015%, latanoprost 0.005% with BAK 0.2mg/ml or latanoprost 0.005%.
* Untreated patients with ocular hypertension must be treatment naïve for the pathology.
* No presence or history of previous ocular diseases other than glaucoma or ocular hypertension, started before the use of hypotensive medication.

Exclusion Criteria:

* Ocular surgery in the previous 6 months.
* Any ocular surface disease not related to inclusion criteria or related issues active within the last 6 months.
* Any topical treatment other than the evaluated in this study in the last 3 months.
* In case of artificial teardrops use, only non conservative ones are allowed, with no more than 4 times per day use, and treatment must be suspended 5 days before inclusion.
* Use of contact lenses in the las 4 weeks.
* Any mental or physical disease that may prevent performing the required tests for the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with ocular hypertension or primary open angle glaucoma
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Inflammatory response in ocular surface secondary to prostaglandin use | 24 hours
  Presence of inflammatory cytokines in ocular surface
Conjunctival cell phenotype and inflammatory infiltration | 24 hours
  Conjunctival cell phenotype assessment by conjunctival in vivo confocal microscopy
Changes in oxidative stress in the tear film | 24 hours
  Changes in oxidative stress at conjunctiva secondary to prostaglandin treatment

CONTACTS AND LOCATIONS:
Locations (1):
- IOBA, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No